CLINICAL TRIAL: NCT01734889
Title: Taste and Palatability of Orfadin Suspension. An Open, Non-controlled 3 Day Study in Pediatric Patients With Hereditary Tyrosinemia Type 1 Treated With Orfadin.
Brief Title: Taste and Palatability of Orfadin Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.NTBC-002
Record Dates: First submitted 2012-11-22; First posted 2012-11-28 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Hereditary Tyrosinemia, Type I
Keywords: nitisinone; Orfadin; suspension; taste; acceptability
MeSH Terms: conditions — Tyrosinemias | interventions — nitisinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Orfadin suspension (Experimental): Drug: nitisinone, oral suspension
  Interventions: Drug: Nitisinone

INTERVENTIONS:
Drug: Nitisinone — Oral suspension

SUMMARY:
The purpose of this study is to verify that pediatric patients, especially those who are not old enough to swallow capsules, accept the taste and palatability of a new suspension.

DETAILED DESCRIPTION:
This is an open, non-randomized, non-controlled, multiple-dose study in 18 pediatric patients. The treatment period is three days, and during the study the subjects will rate the taste and palatability of the suspension or (for younger children) their parents will rate the child´s acceptance of the suspension.

The study consists of a screening period, a 3 day treatment period and a 1 week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HT-1 currently managed on Orfadin (nitisinone) capsules.
* Age from 1 month to less than 18 years.
* Signed informed consent.

Exclusion Criteria:

* Any medical condition which in the opinion of the investigator makes the subject unsuitable for inclusion.
* Enrollment in another concurrent clinical study, or intake of an investigational medicinal product (IMP), within one month prior to inclusion in this study.
* Foreseeable inability to cooperate with given instructions or study procedures.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Brouwer, MD, Study Director — Swedish Orphan Biovitrum
Locations (7):
- Hopital Necker, Paris, France
- Germany (3):
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum der Universität München, München
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Evelina Children's Hospital, St Thomas' Hospital, London
  - St Mary's Hospital, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruitment was performed at seven medical clinics in three countries (United Kingdom, Germany and France). First subject was enrolled on 09 November 2012 and last subject´s last visit was on 01 March 2013.
Groups:
- Orfadin Suspension: Drug: nitisinone, oral suspension 4 mg/mL, twice daily dosing, total daily dose according to current prescribed dose at screening
Period: Overall Study
Arm/Group | Orfadin Suspension
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Orfadin Suspension
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.03 (5.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Region of Enrollment [Number; unit: participants]
  France | 2
  Germany | 4
  United Kingdom | 12

OUTCOME MEASURES:

1. Primary Outcome: The Taste Score for the Last Dose of the Suspension on Day 3 for Subjects 5 - <18 Years
Description: Patients rated the taste of the suspension. The following grading was applied: 5 (very good taste), 4 (good taste), 3 (neither good nor bad taste), 2 (bad taste) and 1 (very bad taste).
Time Frame: Day 3
Population: Full analysis set: All subjects who received at least one dose of study drug and had at least one taste or acceptability assessments
Measure: Median (Full Range); unit: units on a scale
Groups:
- Age 5-<18 Years: Drug: nitisinone, oral suspension 4 mg/mL, twice daily dosing, total daily dose according to current prescribed dose at screening
Arm/Group | Age 5-<18 Years
Number analyzed (Participants) | 12
units on a scale | 4.0 [2.0 to 5.0]

2. Primary Outcome: The Acceptability Score for the Last Dose of the Suspension on Day 3 for Subjects < 5 Years
Description: The parents of patients aged <5 years rated their child´s acceptability of the suspension. The following grading was applied: 5 (very well), 4 (well), 3 (neither well nor badly), 2 (badly) and 1 (very badly).
Time Frame: Day 3
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Groups:
- Age <5 Years: Drug: nitisinone, oral suspension 4 mg/mL, twice daily dosing, total daily dose according to current prescribed dose at screening
Arm/Group | Age <5 Years
Number analyzed (Participants) | 6
units on a scale | 5.0 [4.0 to 5.0]

3. Secondary Outcome: The Palatability Scores on Day 1 (Subjects 5 - < 18 Years)
Description: Patients rated the palatability of the suspension. The following grading was applied: 5 (very good), 4 (good), 3 (neither good nor bad), 2 (bad) and 1 (very bad).
Time Frame: Day 1
Population: Full analysis set: All subjects who received at least one dose of study drug and had at least taste or acceptability assessment.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Age 5-<18 Years
Number analyzed (Participants) | 12
units on a scale | 4.0 [3.0 to 5.0]

4. Secondary Outcome: The Palatability Scores on Day 2 (Subjects 5 - < 18 Years)
Description: as for outcome 3
Time Frame: Day 2
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Age 5-<18 Years
Number analyzed (Participants) | 12
units on a scale | 4.0 [2.0 to 5.0]

5. Secondary Outcome: The Palatability Scores on Day 3 (Subjects 5 - < 18 Years)
Description: as for outcome 3
Time Frame: Day 3
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Age 5-<18 Years
Number analyzed (Participants) | 12
units on a scale | 4.0 [2.0 to 5.0]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded upon administration of first dose until last study visit 1 week after last dose. Serious Adverse Events were recorded from subject signed informed consent until 28 days after last dose.
Arm/Group | Orfadin Suspension
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orfadin Suspension (N=18)
Nasopharyngitis (Infections and infestations) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results are intended to be published as a whole. If no comprehensive publication appears within 12 months of the trial termination, Investigators have the right to publish their results. Such data to be submitted to the Sponsor for review at least 60 days prior to submission for publication, public dissemination, or review by a publication committee. The Sponsor shall be entitled to make a reasoned request that publication be delayed for a period of up to 6 months.